CLINICAL TRIAL: NCT04377048
Title: Nivolumab as add-on to Gemcitabine/S-1 in Metastatic Pancreatic Cancer: a Phase II Trial
Brief Title: Nivolumab Adding on Gemcitabine/S-1 in Metastatic Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry); ACT Genomics (Industry); TTY Biopharm (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202001045MIPA
Record Dates: First submitted 2020-05-04; First posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Stage IV Pancreatic Cancer
Keywords: pancreatic adenocarcinoma; chemotherapy; nivolumab
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Nivolumab; Gemcitabine; tegafur-gimeracil-oteracil; S 1 (combination)

STUDY DESIGN:
Intervention Model Description: Simon's two-stage design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nivolumab/GS (Experimental): Part-1: GS Induction
  * Patients will receive GS for 1 cycle.
  * S-1: 60/80/100 mg per day (based on body surface area, BSA); D1-12; 3 weeks per cycle
  * BSA < 1.25 m2: 60 mg/day; 1.25 m2 ≤ BSA < 1.5 m2: 80 mg/day; BSA ≥ 1.5 m2: 100 mg/day
  * Gemcitabine: 850 mg/m2; D1, 8; 3 weeks per cycle
  * After GS, patients fulfilling the pre-defined CA 19-9 criteria will enter the Add-On part.
  Part-2: Nivolumab Add-On
  * Nivolumab: 3 mg/kg every 2 weeks, 6 weeks per cycle
  * S-1: according to the individualized dose on D8 of cycle 1 in Part-1, 6 weeks per cycle
  * Gemcitabine: according to the individualized dose on D8 of cycle 1 in Part-1, 6 weeks per cycle
  The treatment will be continued until disease progression, intolerance to study treatment or death.
  Interventions: Drug: Nivolumab; Drug: Gemcitabine; Drug: Tegafur-Gimeracil-Oteracil

INTERVENTIONS:
Drug: Nivolumab — as described in "NGS Arm"
Drug: Gemcitabine — as described in "NGS Arm"
Drug: Tegafur-Gimeracil-Oteracil — as described in "NGS Arm"
  Other Names: S-1

SUMMARY:
This study assumes that to achieve significant therapeutic efficacy in advanced pancreatic cancer with immunotherapy, the immune system must remain relatively intact. Therefore, early use, low tumor load, adequate organ function, and slow growth of the tumor are the key points. Stage IV pancreatic adenocarcinoma patients with limited metastatic lesions and adequate organ function will be enrolled. Gemcitabine plus S-1 (GS) will be administered initially, and then CA 19-9 will be evaluated. Those fulfilling pre-defined criteria of CA 19-9 will receive nivolumab add-on therapy.

ELIGIBILITY:
Inclusion Criteria:

1. histologically proven pancreatic adenocarcinoma
2. newly diagnosed, stage IV pancreatic cancer with limited metastases and tumor burden
3. no previous radiotherapy, chemotherapy, targeted therapy, curative surgery, local therapy (eg. radiofrequency ablation, irreversible electroporation, etc.), immunotherapy, cell therapy (autologous or allogenic) used for pancreatic cancer
4. presence of at least one measurable lesion at the pancreas and at least one measurable metastatic lesion
5. age between 20 and 75 years at registration
6. ECOG performance status of 0 or 1
7. adequate major organ functions
8. baseline CA 19-9 > upper limit of normal
9. Glasgow prognostic score of 0 (ie. albumin ≥ 3.5 g/dL and CRP ≤ 1 mg/dL)
10. ability to take study medication (S-1) orally
11. no clinically significant abnormal ECG findings within 28 days prior to registration
12. Women of childbearing potential (including women with chemical menopause or no menstruation for other medical reasons) must agree to use contraception from the time of informed consent until 5 months or more after the last dose of investigational products. Also, women must agree not to breastfeed from the time of informed consent until 5 months or more after the last dose of the investigational product.
13. Men must agree to use contraception from the start of study treatment until 7 months or more after the last dose of the investigational product.
14. Sign written informed consent

Exclusion Criteria:

1. interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected treatment-related pulmonary toxicity within 28 days prior to registration
2. presence of diarrhea ≥ CTCAE v.5.0 grade 2
3. concomitant systemic infection requiring treatment
4. clinically significant co-morbid medical conditions, including cardiovascular disease known autoimmune disease
5. concurrent autoimmune disease or history of chronic or recurrent autoimmune disease
6. prior organ allograft or allogeneic bone marrow transplantation
7. received systemic corticosteroids (except for temporary use, e.g., for examination or prophylaxis of allergic reactions) or immunosuppressants within 28 days before registration
8. HBV (positive HBsAg or HBV DNA) or HCV carrier (positive anti-HCV or HCV RNA)
9. known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome
10. moderate or severe ascites, pleural effusion, or pericardial effusion requiring treatment
11. central nervous system metastasis
12. prior or concurrent malignancies within the last 3 years, with the exception of carcinoma in situ of the cervix, or basal type skin cancer
13. concomitant treatment with flucytosine, phenytoin or warfarin
14. any major surgery within 4 weeks of study treatment. Participants must have recovered from the effects of major surgery or significant traumatic injury at least 14 days before the first dose of study treatment.
15. transfusion from 72 hours prior to registration to the first dose of study drug administration
16. pregnant women or nursing mothers, or positive pregnancy tests
17. severe mental disorder
18. treatment with botanical preparations (eg, herbal supplements or traditional Chinese medicines) intended for general health support or to treat the disease under study within 2 weeks prior to registration
19. vaccine therapies for prevention of infectious diseases within 4 weeks of study drug administration except inactivated seasonal influenza vaccine
20. any condition requiring anti-platelet or anticoagulant therapy within 12 weeks prior to registration
21. oral or iv antibiotic use within 2 weeks prior to registration
22. uncontrollable pain caused by a tumor
23. receiving antineoplastic agents within 28 days before registration
24. patients judged by the principal investigator or subinvestigators to be inappropriate as subjects of this study

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
response rate | 6 weeks
  overall response rate of gemcitabine/S-1/nivolumab

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Hung Yang, M.D., Ph.D., Principal Investigator — Department of Oncology, National Taiwan University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ueno H, Ioka T, Ikeda M, Ohkawa S, Yanagimoto H, Boku N, Fukutomi A, Sugimori K, Baba H, Yamao K, Shimamura T, Sho M, Kitano M, Cheng AL, Mizumoto K, Chen JS, Furuse J, Funakoshi A, Hatori T, Yamaguchi T, Egawa S, Sato A, Ohashi Y, Okusaka T, Tanaka M. Randomized phase III study of gemcitabine plus S-1, S-1 alone, or gemcitabine alone in patients with locally advanced and metastatic pancreatic cancer in Japan and Taiwan: GEST study. J Clin Oncol. 2013 May 1;31(13):1640-8. doi: 10.1200/JCO.2012.43.3680. Epub 2013 Apr 1. PMID 23547081
- [Result] Weiss GJ, Blaydorn L, Beck J, Bornemann-Kolatzki K, Urnovitz H, Schutz E, Khemka V. Phase Ib/II study of gemcitabine, nab-paclitaxel, and pembrolizumab in metastatic pancreatic adenocarcinoma. Invest New Drugs. 2018 Feb;36(1):96-102. doi: 10.1007/s10637-017-0525-1. Epub 2017 Nov 8. PMID 29119276
- [Derived] Yang SH, Chen BB, Lee JC, Kuo YT, Kuo SH, Cheng AL, Yeh KH. Incorporating nivolumab with preceded gemcitabine and S-1 chemotherapy for patients of metastatic pancreatic cancer: a pilot study. Am J Cancer Res. 2025 Sep 25;15(9):4108-4120. doi: 10.62347/NJOX8790. eCollection 2025. PMID 41113977